CLINICAL TRIAL: NCT01481792
Title: Use of the VisuMax Femtosecond Laser for the Correction of Myopia With Small Incision Lenticular Extraction
Brief Title: Efficacy and Safety of ReLEx Smile for Laser Correction of Myopia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Jesper Hjortdal, Professor, consultant, MD, PhD, University of Aarhus
Other Study IDs: AUH-Ophthalmology-2011-01
Record Dates: First submitted 2011-11-23; First posted 2011-11-30 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Myopia
Keywords: Keratorefractive Surgical Procedures
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the safety and efficacy of the Carl Zeiss Meditec VisuMax femtosecond laser for lamellar resection (ReLEx smile) in the reduction of myopia.

DETAILED DESCRIPTION:
Quality control study of patients treated with ReLEx smile for myopia at the Department of Ophthalmology, Aarhus University Hospital.

The patients will be followed with standard clinical techniques (slit-lamp examination, refraction, topography) during their normal follow-up up to 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Indication for keratorefractive correction of myopia
* Patient consent to undergo keratorefractive correction of myopia

Exclusion Criteria:

* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Department of Ophthalmology, Aarhus University Hospital, for keratorefractive surgical correction of myopia
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Refraction one year after surgery
  Achieved change in refraction (spherical equivalent, SE) in diopters will be compared with attempted change in refraction (SE) in diopters. Data will be reported as fraction of eyes within an error (achieved - attempted) of +/- 0.5 diopters (SE) and within an error of +/- 1 diopters (SE).
Safety | One year after surgery
  Data will be reported as:
  * Percentage of eyes with best spectacle corrected visual acuity (BSCVA) worse than 20/40 for eyes with BSCVA of 20/20 or better before survey
  * Percentage of eyes that lose 2 Snellen lines or more of BSCVA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Aarhus University Hospital, Aarhus C, Denmark